CLINICAL TRIAL: NCT06154122
Title: The Feasibility of Virtual Reality-Based Activities for Upper Limb Rehabilitation of People With Acute/Sub-Acute Tetraplegia
Brief Title: Virtual Reality Upper Limb Therapy for People With Spinal Cord Injury
Acronym: VRULT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VRULT
Record Dates: First submitted 2023-11-02; First posted 2023-12-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Tetraplegia; Spinal Cord Injuries; Upper Extremity Paralysis
Keywords: Virtual Reality; Upper Extremities; Acute/Sub-acute Rehabilitation
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Plus Treatment As Usual (Experimental): 3 sessions of virtual reality upper limb treatment for up to 30 minutes each will be administered each week for 12 weeks.
  Participants randomised to the VR treatment arm will also receive treatment as usual for their upper limbs (see Treatment As Usual).
  Interventions: Device: Virtual Reality Upper Limb Rehabilitation Games; Other: Upper Limb Rehabilitation
- Treatment As Usual (Active Comparator): Usual upper limb rehabilitation is delivered by occupational therapists and physiotherapists and aims to build strength of the upper limbs and optimise function. Patients receive hand therapy once per day and physiotherapy twice per day. Rehabilitation is highly individualised.
  Interventions: Other: Upper Limb Rehabilitation

INTERVENTIONS:
Device: Virtual Reality Upper Limb Rehabilitation Games — A VR upper limb rehabilitation programme prescribed by the therapist with games chosen depending on the exercise task required and the level of difficulty adapted to the ability of the individual. The participant will use the VR system's user interface to navigate through menus to set their gameplay preferences and select which games to play.
  The games of the intervention will involve facilitating and replicating upper limb movements including gross movements of the shoulder, such as rotation, abduction and addiction, movements of the upper and lower arms, such as flexion and extension of the elbow, and hand, wrist and finger movements, including wrist pronation supination, and finger flexion and extension, as well as tenodesis movements, grasping, and pinching.
  Arms: Virtual Reality Plus Treatment As Usual
Other: Upper Limb Rehabilitation — Usual upper limb rehabilitation is delivered by occupational therapists and physiotherapists and aims to build strength of the upper limbs and optimise function. Patients receive hand therapy once per day and physiotherapy twice per day. Rehabilitation is highly individualised.

SUMMARY:
This study aims to test if the VR games could be a form of upper limb rehabilitation for people with arm/hand problems due to SCI while they are in hospital. Participants who have had a spinal cord injury and have tetraplegia will be recruited from the Queen Elizabeth National Spinal Injuries Unit. After they have provided informed consent, they will receive 12 weeks of either standard upper limb therapy ('control group'), or both the VR activities and standard treatment ('VR Group'). Participants who receive VR activities will engage in immersive VR games that have been designed in co-production with people with tetraplegia and spinal cord injury specialists. The games aim to help participants improve the use of their arms and hands while they are undergoing primary rehabilitation within the Queen Elizabeth National Spinal Injuries Unit (QENSIU). The participants who are in the control group will receive their usual rehabilitation and will be given the opportunity to try the VR games after the completion of their involvement in the trial.

This study will measure the feasibility (the 'primary outcome') and explore the effectiveness (the 'secondary outcome') of the VR intervention. Feasibility will be measured by recording how often the VR games are used and whether or not participants use the games for the full duration of the trial. Participants and therapists will be interviewed at the end of the trial.

DETAILED DESCRIPTION:
A spinal cord injury (SCI) impacts nearly every aspect of a person's life. People with SCI will have muscular paralysis and loss of sensory and autonomic function below the level of their injury. Immediately following injury, people with SCI require acute in-patient care, during which rehabilitation is started. Following an SCI, people are at risk of pressure ulcers, urinary tract infections, spasticity, autonomic dysreflexia, depression, neuropathic pain, difficulty breathing, and circulatory problems. The multitude of impairments following SCI are associated with lower quality of life.

Reducing reliance on care and achieving higher levels of independence is a major goal for people with SCI. People with SCI can improve the motor power and therefore function of their paralysed limbs through rehabilitation. This enables people with SCI to carry out tasks which would otherwise require a carer. Dressing, bladder and bowel care, transferring in and out of a wheelchair, and feeding are activities that often require more assistance. The difficulty in carrying out these activities can be greatly reduced if people with SCI can recover function in the upper limbs. Even small improvements in limb function can have large effects on a people with SCI's independence.

For people with tetraplegia, where the injury affects all four limbs, improving upper limb function is a major focus of rehabilitation. People with tetraplegia reported improvement in hand and arm function as their highest priority for improvement compared to other rehabilitation targets. Improvements in upper limb function can be achieved through Activity-Based Therapy (ABT). ABT refers to any intervention that involves high intensity, repetitive exercises which target activity-dependent plasticity in spinal circuits. The improvements from ABT in upper limb function have greater effects on quality of life when compared to traditional physical interventions targeted above the level of injury. Exercise can alleviate symptoms of some secondary conditions which can positively impact on quality of life. Physical inactivity is often reported by spinal cord injured people, with limited access to exercise being just one of many barriers to active lifestyles. There is a clear need to improve the accessibility of therapy for people with SCI.

Virtual Reality (VR) technology used as an assistive device for upper limb rehabilitation has good potential for people with SCI during rehabilitation by facilitating greater adherence to therapy and increasing access to the most effective rehabilitation strategies for people with neurological disorders. However, currently only a few studies have investigated the use of VR in SCI rehabilitation of the upper limbs. Of these studies, most have reported positive outcomes.

Three systematic reviews on the use of VR after spinal cord injury have been published in the last few years. Overall the findings suggest that VR training can improve motor function and balance, reduce symptoms such as pain, and improve aerobic function. However, there were consistent limitations reported including a relatively small number of studies, small experimental samples, and no consensus on the optimal treatment parameters or technology employed. Furthermore, there were no studies that evaluated the use of VR in the acute phase following SCI when there is most potential for recovery.

VR can have positive psychological effects among people with an SCI such as increased self-confidence, motivation, and participation in therapy. ABT has been shown to improve function through neuromuscular recovery and increase participation in therapy. The principles of ABT which target motor improvement could be integrated into a VR intervention for upper limb rehabilitation, which could provide a promising and exciting option for people with SCI in early stages of recovery.

There are challenges in the delivery of ABT, such as the cost associated with using assistive devices, resources required to train staff, difficulty achieving sufficient dosage, factors such as motivation to engage in therapy, and access to therapy equipment. These challenges could be overcome by collaborating with people with SCI and their carers at the design stage of an intervention to impart valuable expertise about their chronic conditions, experiences of the acute phase recovery immediately following injury, and ideas about how to better manage rehabilitation. This intervention has been developed using co-production, where end-users (people with SCI and SCI therapists) were involved at every stage of the development process. This process can produce interventions that are highly accepted and efficacious.

The investigators have therefore developed a set of VR-based physical exercises for upper limb rehabilitation in collaboration with people with lived experience of tetraplegia and spinal cord injury specialists. VR will allow the participant to repeatedly experience engaging, fun, and motivating digital environments within which can be practised upper limb movements as an adjunct to standard upper limb rehabilitation. The aim of this randomised controlled feasibility study is to determine if this intervention is usable and acceptable for people with tetraplegia and therapists during acute rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial.
* Aged 18 years or above.
* An in-patient at the Queen Elizabeth National Spinal Injuries Unit in Glasgow with a diagnosis of tetraplegia.
* Sustained a cervical spine injury (C4-C8).
* Medically stable to engage in physical rehabilitation and physical activity.
* Sitting up in a wheelchair for at least 2 hours daily.

Exclusion Criteria:

* Scheduled elective surgery or other procedures requiring general anaesthesia anticipated within the next 12 weeks.
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participated in another research trial involving an investigational product in the past 12 weeks.
* Participating in another research trial investigating upper limb rehabilitation interventions.
* Self-reported motion sickness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Number of VR Sessions Completed | Measured over 12 weeks of participation.
  The number of sessions of VR the participant completes. This will be recorded as an integer value from 0 to 3 per week of participation.
Time spent in VR | Measured over 12 weeks of participation.
  The time spent using the VR games, as recorded by the device. This will be measured in minutes and seconds.
Number of completed assessments | Measured over 12 weeks of participation.
  Completion of the assessments used at baseline, midpoint, and endpoint of the study.
Participant retention | Measured over 12 weeks of participation.
  The number of participants recruited to the study per month will be combined with eligibility and retention to determine overall recruitment and retention.
Participant recruitment rate per month | Measured over 12 weeks of participation.
  The number of participants recruited to the study per month will be combined with eligibility and retention to determine overall recruitment and retention.
Participant eligibility | Measured over 12 weeks of participation.
  Number of people approached about the study and the number of people who meet the inclusion and exclusion criteria.
  The number of participants recruited to the study per month will be combined with eligibility and retention to determine overall recruitment and retention.
Adverse event monitoring and reporting | Measured over 12 weeks of participation.
  Monitoring and reporting of any adverse events, either during or immediately following the VR intervention will be combined with results from semi-structured interviews and questionnaires to determine acceptability and usability.
Semi-structured Interviews | Completed at week 12 after the last VR session has been completed.
  Determine the usability of the intervention through semi-structured interviews with participants and therapists.
  Monitoring and reporting of any adverse events, either during or immediately following the VR intervention will be combined with results from semi-structured interviews and questionnaires to determine acceptability and usability.
Usefulness, Satisfaction, and Ease of use Questionnaire (USE Questionnaire) | Completed at week 12 after the last VR session has been completed.
  Determine the usability of the intervention through questionnaire with participants and therapists (USE Questionnaire (Lund 2001)). This a 30-item survey.
  The maximum value for the USE Questionnaire is 210, and the minimum is 7. Participants can also respond 'not applicable' to all items.
  Higher scores mean a better outcome. Individual subscores of the USE Questionnaire can indicate that the system is or is not useful, satisfying, and/or easy to use.
Handedness (Treatment Parameter) | Completed at week 12 after the last VR session has been completed.
  The participant's choice of left, right, or both arm(s)/hand(s) will be recorded per session.
  Recording the treatment parameters the participant using VR selects during therapy to determine usability in combination with the interviews and questionnaires.
Target Movement (Treatment Parameters) | Completed at week 12 after the last VR session has been completed.
  The participant's choice of the type of movement they want to practise will be recorded per session. Movements will include wrist pronation/supination, elbow flexion/extension, and an integrated movement incorporating shoulder movement and elbow flexion and extension.
  Recording the treatment parameters the participant using VR selects during therapy to determine usability in combination with the interviews and questionnaires.
Number of Repetitions (Treatment Parameters) | Completed at week 12 after the last VR session has been completed.
  The number of repetitions of the target movement (see outcome 11) will be recorded per session.
  Recording the treatment parameters the participant using VR selects during therapy to determine usability in combination with the interviews and questionnaires.
Choice of Game (Treatment Parameters) | Completed at week 12 after the last VR session has been completed.
  The participant's choice of game will be recorded per session.
  Recording the treatment parameters the participant using VR selects during therapy to determine usability in combination with the interviews and questionnaires.
Input Device choices (Treatment Parameters) | Completed at week 12 after the last VR session has been completed.
  The participant's choice of input device will be recorded per session. Input devices available will include either the use of tracked hand-held controllers, or the use of an infrared-based 'hand-held controller-free' hand-tracking module.
  Recording the treatment parameters the participant using VR selects during therapy to determine usability in combination with the interviews and questionnaires.

SECONDARY OUTCOMES:
Motor Score | Measured at baseline, 6 weeks, and 12 weeks.
  Explore effectiveness of the VR-based upper limb rehabilitation intervention for people with tetraplegia during the acute, in-patient stage of rehabilitation.
  Higher scores on the motor score indicate a better outcome, ranging between 0 and 50.
  i. Motor score using the Upper Extremity Motor Score (UEMS) (Rupp et al., 2021).
  Motor score, sensation, independence, hand/upper limb function, and pain measures will be use to explore effectiveness.
Sensation | Measured at baseline, 6 weeks, and 12 weeks.
  Explore effectiveness of the VR-based upper limb rehabilitation intervention for people with tetraplegia during the acute, in-patient stage of rehabilitation.
  Higher scores on the light touch and pin prick scale indicate better outcomes, ranging between 0 and 112.
  ii. Sensation (assess light touch and pin prick according to the ISNCSCI) (Rupp et al., 2021).
  Motor score, sensation, independence, hand/upper limb function, and pain measures will be use to explore effectiveness.
Independence | Measured at baseline, 6 weeks, and 12 weeks.
  Explore effectiveness of the VR-based upper limb rehabilitation intervention for people with tetraplegia during the acute, in-patient stage of rehabilitation.
  iii. Independence evaluated by the Spinal Cord Independence Measure (SCIM-III) (Itzkovich et al., 2007).
  There are a total of 19 items on the SCIM III, which are divided into 3 subscales (self-care, respiration and sphincter management, and mobility). A total score out of 100 is achieved, with the subscales weighted as follows: self-care: scored 0-20; respiration and sphincter management: scored 0-40; and mobility: scored 0-40. Scores are higher in patients that require less assistance or fewer aids to complete basic activities of daily living and life support activities.
  Motor score, sensation, independence, hand/upper limb function, and pain measures will be use to explore effectiveness.
Hand/Upper Limb Function | Measured at baseline, 6 weeks, and 12 weeks.
  iv. Hand/Upper Limb Function by the Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) Subscales (Kalsi-Ryan et al., 2012).
  Subtests of the GRASSP include manual muscle testing (which is graded on a scale of 0-5 for each selected muscle, with higher values representing greater muscle strength), sensation testing (which is graded on a scale of 0-4 for 3 areas, with higher scores representing greater sensation), prehension ability (which is scored on a scale of 0-4 for 3 grasp patterns with higher scores representing better ability to perform grasp with normal strength), and prehension performance (which is graded on a score of 0-5 for 4 different tasks, with higher scores representing better hand function).
Pain Intensity | Measured at baseline, 6 weeks, and 12 weeks.
  Explore effectiveness of the VR-based upper limb rehabilitation intervention for people with tetraplegia during the acute, in-patient stage of rehabilitation.
  v. Pain measured on a Visual Analogue Scale.
  A Visual Analogue Scale will be shown to participants, which is a 10 cm-long horizontal like with indices ranging from 0 to 10. The participant marks their current pain along the line. Higher scores represent a worse outcome, indicating higher pain at that specific timepoint.
  Motor score, sensation, independence, hand/upper limb function, and pain measures will be use to explore effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Paul, PhD, Principal Investigator — Glasgow Caledonian University; Matthieu Poyade, PhD, Study Chair — Glasgow School of Art
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit (NHS Greater Glasgow and Clyde), Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publications will be available at request to other researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be stored on One Drive for 5 years, after which it will be deleted and CRFs will be shredded as confidential waste.
Access Criteria: All IPD that underlie results in a publication will be available at request and stored on a Glasgow Caledonian University OneDrive account.

REFERENCES:
- [Background] Adriaansen JJ, Ruijs LE, van Koppenhagen CF, van Asbeck FW, Snoek GJ, van Kuppevelt D, Visser-Meily JM, Post MW. Secondary health conditions and quality of life in persons living with spinal cord injury for at least ten years. J Rehabil Med. 2016 Nov 11;48(10):853-860. doi: 10.2340/16501977-2166. PMID 27834436
- [Background] van den Akker LE, Holla JFM, Dadema T, Visser B, Valent LJ, de Groot S, Dallinga JM, Deutekom M; WHEELS-study group. Determinants of physical activity in wheelchair users with spinal cord injury or lower limb amputation: perspectives of rehabilitation professionals and wheelchair users. Disabil Rehabil. 2020 Jul;42(14):1934-1941. doi: 10.1080/09638288.2019.1577503. Epub 2019 Mar 29. PMID 30924706
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Anderson KD. Equitable partnerships between scientists and persons living with spinal cord injury will strengthen research scope, quality, and outcomes. Curr Opin Neurol. 2021 Dec 1;34(6):783-788. doi: 10.1097/WCO.0000000000000989. PMID 34545013
- [Background] de Araujo AVL, Neiva JFO, Monteiro CBM, Magalhaes FH. Efficacy of Virtual Reality Rehabilitation after Spinal Cord Injury: A Systematic Review. Biomed Res Int. 2019 Nov 13;2019:7106951. doi: 10.1155/2019/7106951. eCollection 2019. PMID 31828120
- [Background] Behrman AL, Ardolino EM, Harkema SJ. Activity-Based Therapy: From Basic Science to Clinical Application for Recovery After Spinal Cord Injury. J Neurol Phys Ther. 2017 Jul;41 Suppl 3(Suppl 3 IV STEP Spec Iss):S39-S45. doi: 10.1097/NPT.0000000000000184. PMID 28628595
- [Background] Bickenbach, J. et al. (2013) 'Chapter 4: Health care and rehabilitation needs.', in International perspectives on spinal cord injury / edited by Jerome Bickenbach. Geneva: World Health Organization, pp. 67-91.
- [Background] Bryce TN, Budh CN, Cardenas DD, Dijkers M, Felix ER, Finnerup NB, Kennedy P, Lundeberg T, Richards JS, Rintala DH, Siddall P, Widerstrom-Noga E. Pain after spinal cord injury: an evidence-based review for clinical practice and research. Report of the National Institute on Disability and Rehabilitation Research Spinal Cord Injury Measures meeting. J Spinal Cord Med. 2007;30(5):421-40. doi: 10.1080/10790268.2007.11753405. PMID 18092558
- [Background] Buchholz AC, Martin Ginis KA, Bray SR, Craven BC, Hicks AL, Hayes KC, Latimer AE, McColl MA, Potter PJ, Wolfe DL. Greater daily leisure time physical activity is associated with lower chronic disease risk in adults with spinal cord injury. Appl Physiol Nutr Metab. 2009 Aug;34(4):640-7. doi: 10.1139/H09-050. PMID 19767799
- [Background] Cragg J, Krassioukov A. Autonomic dysreflexia. CMAJ. 2012 Jan 10;184(1):66. doi: 10.1503/cmaj.110859. Epub 2011 Oct 11. No abstract available. PMID 21989470
- [Background] De Miguel-Rubio A, Rubio MD, Salazar A, Camacho R, Lucena-Anton D. Effectiveness of Virtual Reality on Functional Performance after Spinal Cord Injury: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2020 Jul 1;9(7):2065. doi: 10.3390/jcm9072065. PMID 32630234
- [Background] Filipcic T, Sember V, Pajek M, Jerman J. Quality of Life and Physical Activity of Persons with Spinal Cord Injury. Int J Environ Res Public Health. 2021 Aug 30;18(17):9148. doi: 10.3390/ijerph18179148. PMID 34501739
- [Background] Gao, M., Kortum, P. and Oswald, F. (2018) 'Psychometric Evaluation of the USE (Usefulness, Satisfaction, and Ease of use) Questionnaire for Reliability and Validity', Proceedings of the Human Factors and Ergonomics Society Annual Meeting, 62(1), pp. 1414-1418. Available at: https://doi.org/10.1177/1541931218621322.
- [Background] Hoekstra F, Gainforth HL, Broeksteeg R, Corras S, Collins D, Gaudet S, Giroux EE, McCallum S, Ma JK, Rakiecki D, Rockall S, van den Berg-Emons R, van Vilsteren A, Wilroy J, Martin Ginis KA. Theory- and evidence-based best practices for physical activity counseling for adults with spinal cord injury. J Spinal Cord Med. 2024 Jul;47(4):584-596. doi: 10.1080/10790268.2023.2169062. Epub 2023 Mar 29. PMID 36988416
- [Background] Itzkovich M, Gelernter I, Biering-Sorensen F, Weeks C, Laramee MT, Craven BC, Tonack M, Hitzig SL, Glaser E, Zeilig G, Aito S, Scivoletto G, Mecci M, Chadwick RJ, El Masry WS, Osman A, Glass CA, Silva P, Soni BM, Gardner BP, Savic G, Bergstrom EM, Bluvshtein V, Ronen J, Catz A. The Spinal Cord Independence Measure (SCIM) version III: reliability and validity in a multi-center international study. Disabil Rehabil. 2007 Dec 30;29(24):1926-33. doi: 10.1080/09638280601046302. Epub 2007 Mar 5. PMID 17852230
- [Background] Jervis Rademeyer H, Gauthier C, Zariffa J, Walden K, Jeji T, McCullum S, Musselman KE. Using activity-based therapy for individuals with spinal cord injury or disease: Interviews with physical and occupational therapists in rehabilitation hospitals. J Spinal Cord Med. 2023 Mar;46(2):298-308. doi: 10.1080/10790268.2022.2039855. Epub 2022 Mar 29. PMID 35349399
- [Background] Kalsi-Ryan S, Beaton D, Curt A, Duff S, Popovic MR, Rudhe C, Fehlings MG, Verrier MC. The Graded Redefined Assessment of Strength Sensibility and Prehension: reliability and validity. J Neurotrauma. 2012 Mar 20;29(5):905-14. doi: 10.1089/neu.2010.1504. Epub 2011 Aug 12. PMID 21568688
- [Background] Kalsi-Ryan S, Beaton D, Ahn H, Askes H, Drew B, Curt A, Popovic MR, Wang J, Verrier MC, Fehlings MG. Responsiveness, Sensitivity, and Minimally Detectable Difference of the Graded and Redefined Assessment of Strength, Sensibility, and Prehension, Version 1.0. J Neurotrauma. 2016 Feb 1;33(3):307-14. doi: 10.1089/neu.2015.4217. Epub 2015 Dec 17. PMID 26560017
- [Background] Kazim SF, Bowers CA, Cole CD, Varela S, Karimov Z, Martinez E, Ogulnick JV, Schmidt MH. Corticospinal Motor Circuit Plasticity After Spinal Cord Injury: Harnessing Neuroplasticity to Improve Functional Outcomes. Mol Neurobiol. 2021 Nov;58(11):5494-5516. doi: 10.1007/s12035-021-02484-w. Epub 2021 Aug 3. PMID 34341881
- [Background] Kramer JL, Lammertse DP, Schubert M, Curt A, Steeves JD. Relationship between motor recovery and independence after sensorimotor-complete cervical spinal cord injury. Neurorehabil Neural Repair. 2012 Nov-Dec;26(9):1064-71. doi: 10.1177/1545968312447306. Epub 2012 May 30. PMID 22647878
- [Background] Lewis NE, Tabarestani TQ, Cellini BR, Zhang N, Marrotte EJ, Wang H, Laskowitz DT, Abd-El-Barr MM, Faw TD. Effect of Acute Physical Interventions on Pathophysiology and Recovery After Spinal Cord Injury: A Comprehensive Review of the Literature. Neurospine. 2022 Sep;19(3):671-686. doi: 10.14245/ns.2244476.238. Epub 2022 Sep 30. PMID 36203293
- [Background] Lu X, Battistuzzo CR, Zoghi M, Galea MP. Effects of training on upper limb function after cervical spinal cord injury: a systematic review. Clin Rehabil. 2015 Jan;29(1):3-13. doi: 10.1177/0269215514536411. Epub 2014 Jun 4. PMID 25575932
- [Background] Miguel-Rubio A, Rubio MD, Salazar A, Moral-Munoz JA, Requena F, Camacho R, Lucena-Anton D. Is Virtual Reality Effective for Balance Recovery in Patients with Spinal Cord Injury? A Systematic Review and Meta-Analysis. J Clin Med. 2020 Sep 4;9(9):2861. doi: 10.3390/jcm9092861. PMID 32899665
- [Background] Quel de Oliveira C, Refshauge K, Middleton J, de Jong L, Davis GM. Effects of Activity-Based Therapy Interventions on Mobility, Independence, and Quality of Life for People with Spinal Cord Injuries: A Systematic Review and Meta-Analysis. J Neurotrauma. 2017 May 1;34(9):1726-1743. doi: 10.1089/neu.2016.4558. Epub 2016 Dec 20. PMID 27809702
- [Background] Dolbow DR, Gorgey AS, Recio AC, Stiens SA, Curry AC, Sadowsky CL, Gater DR, Martin R, McDonald JW. Activity-Based Restorative Therapies after Spinal Cord Injury: Inter-institutional conceptions and perceptions. Aging Dis. 2015 Aug 1;6(4):254-61. doi: 10.14336/AD.2014.1105. eCollection 2015 Aug. PMID 26236547
- [Background] Roy RR, Harkema SJ, Edgerton VR. Basic concepts of activity-based interventions for improved recovery of motor function after spinal cord injury. Arch Phys Med Rehabil. 2012 Sep;93(9):1487-97. doi: 10.1016/j.apmr.2012.04.034. PMID 22920448
- [Background] Rupp R, Biering-Sorensen F, Burns SP, Graves DE, Guest J, Jones L, Read MS, Rodriguez GM, Schuld C, Tansey-Md KE, Walden K, Kirshblum S. International Standards for Neurological Classification of Spinal Cord Injury: Revised 2019. Top Spinal Cord Inj Rehabil. 2021 Spring;27(2):1-22. doi: 10.46292/sci2702-1. No abstract available. PMID 34108832
- [Background] Savic G, Frankel HL, Jamous MA, Soni BM, Charlifue S. Participation restriction and assistance needs in people with spinal cord injuries of more than 40 year duration. Spinal Cord Ser Cases. 2018 Mar 27;4:28. doi: 10.1038/s41394-018-0056-9. eCollection 2018. PMID 29619249
- [Background] Schiza E, Matsangidou M, Neokleous K, Pattichis CS. Virtual Reality Applications for Neurological Disease: A Review. Front Robot AI. 2019 Oct 16;6:100. doi: 10.3389/frobt.2019.00100. eCollection 2019. PMID 33501115
- [Background] Slattery P, Saeri AK, Bragge P. Research co-design in health: a rapid overview of reviews. Health Res Policy Syst. 2020 Feb 11;18(1):17. doi: 10.1186/s12961-020-0528-9. PMID 32046728
- [Background] Yeo E, Chau B, Chi B, Ruckle DE, Ta P. Virtual Reality Neurorehabilitation for Mobility in Spinal Cord Injury: A Structured Review. Innov Clin Neurosci. 2019 Jan 1;16(1-2):13-20. PMID 31037223
- See also: Meta (2023) 'Meta Quest 2 Technical Specifications'. Meta Platforms, Inc. Available at: https://www.meta.com/gb/quest/products/quest-2/tech-specs/#tech-specs. — https://www.meta.com/gb/quest/products/quest-2/tech-specs/

DOCUMENTS (1):
  • Study Protocol (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT06154122/Prot_000.pdf